CLINICAL TRIAL: NCT01547806
Title: Mobilization and Collection of Autologous Stem Cell for Transplantation (ASCT) for Plasma Cell Myeloma (PCM)
Brief Title: Collection of Transplant Stem Cells for Plasma Cell Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jennifer Kanakry, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120074; 12-C-0074
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Plasma Cell Myeloma; Multiple Myeloma
Keywords: Autologous Hematopoietic Cell Transplantation; Plasma Cell Myeloma; Mobilization; Apheresis; Plerixafor
MeSH Terms: conditions — Multiple Myeloma | interventions — Filgrastim; plerixafor; Blood Component Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hematopoietic Progenitor Cells (HPC) (Experimental): Subjects will undergo mobilization and collection of HPC, Apheresis for subsequent use in various clinical protocols.
  Interventions: Drug: Filgrastim; Drug: Plerixafor; Procedure: Apheresis

INTERVENTIONS:
Drug: Filgrastim — Filgrastim will be administered as a single daily dose in a dose range of 10-16ug/kg/day subcutaneously for 5-7days
  Other Names: Neupogen
Drug: Plerixafor — Plerixafor will be given on day 4, 8-10 hours before the day 5 apheresis, dose calculated according to patient weight
  Other Names: Mozobil
Procedure: Apheresis — The minimum cluster of differentiation 34 (CD34)+ cell dose that must be collected in order to proceed with a single autologous transplantation is 2 x 106 CD34+ cells/kg.

SUMMARY:
Background:

- One beneficial treatment for plasma cell myeloma is high-dose chemotherapy followed by stem cell transplant. Researchers want to collect stem cells from the blood for later transplant.

Objectives:

- To collect stem cells for transplant as part of treatment for plasma cell myeloma.

Eligibility:

- Individuals at least 18 years of age who will have chemotherapy and stem cell transplant for plasma cell myeloma.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Participants will have filgrastim injections for 5 days before collection. This will move stem cells from the bone marrow to the blood.
* Participants will have apheresis to collect the stem cells.
* Participants who need additional apheresis procedures to collect stem cells will have filgrastim and a dose of plerixafor to improve the collection yield.

DETAILED DESCRIPTION:
Background:

High-dose chemotherapy followed by autologous hematopoietic cell transplant (AHCT) remains a critical part of the Plasma Cell Myeloma (PCM) treatment in subjects eligible for the procedure. The timing of the procedure however, has become more controversial recently. This protocol will allow collection of Hematopoietic Progenitor Cells by Apheresis (HPC, Apheresis) in potential candidates for various PCM protocols at the Clinical Center.

The mobilizing agent plerixafor (Mozobil, Genzyme) has been recently approved by the Food and Drug Administration (FDA) for mobilization in PCM. However, the best and most cost effective strategy for its use remains to be defined.

Objectives:

Evaluate the overall validity of an HPC mobilization strategy (with granulocyte-colony stimulating factor (G-CSF) alone or in combination with plerixafor) using a formula calculating the likelihood of collecting greater than or equal to 5 time 10^6 cluster of differentiation 34 (CD34) plus cells/kg in a single mobilization cycle.

Collect mobilized Hematopoietic Progenitor Cells by Apheresis (HPC, Apheresis) prior to AHCT for PCM

Eligibility:

Subjects with a possible indication for AHCT for the treatment of newly diagnosed PCM.

Subjects with recurrent or persistent evaluable disease who have not undergone AHCT for the treatment of the PCM.

Design:

Subjects will undergo mobilization and collection of HPC, Apheresis for subsequent use in various clinical protocols.

Mobilization will be provided by a 5-daily administration of filgrastim according to standard procedure.

The need for an additional mobilizing agent (plerixafor) to be given on day 4 of mobilization will be evaluated in real time in each patient, based on the peripheral blood CD34 count on the morning of day 4 of filgrastim administration.

Study accrual over a 3-year period: 70 subjects

ELIGIBILITY:
* INCLUSION CRITERIA:

Multiple Myeloma Criteria:

Subjects with an indication for autologous hematopoietic cell transplant (AHCT) for the treatment of PCM as determined by the principal investigator (PI) or lead associate investigator (LAI).

* Subjects following induction treatment for plasma cell myeloma (PCM)
* Subjects with recurrent or persistent evaluable disease who have not undergone AHCT for the treatment of the PCM.

Other Eligibility Criteria:

Age greater than or equal to 18 years and less than or equal to 75 years. In subjects between 65 and 75 years of age, physiologic age and co-morbidity will be thoroughly evaluated before enrolling.

Karnofsky performance status of 70% or greater (Eastern Cooperative Oncology Group ((ECOG) 0 or 1)

Ejection fraction (EF) by multigated acquisition scan (MUGA) or 2-D echocardiogram within institution normal limits. In case of low ejection fraction (EF), the subject may remain eligible after a stress echocardiogram is performed if the EF is more than 35% and if the increase in EF with stress is estimated at 10% or more.

Hemoglobin (Hgb) greater than or equal to 8 g/dl (transfusion acceptable)

No history of abnormal bleeding tendency.

Patients must be able to give informed consent

EXCLUSION CRITERIA:

Prior allogeneic stem cell transplantation

Hypertension not adequately controlled by 3 or less medications.

Clinically significant cardiac pathology: myocardial infarction within 6 months prior to enrollment, Class III or IV heart failure according to New York Heart Association (NYHA), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Specifically, any history of cardio-vascular pathology or symptoms, not clearly fitting this exclusion criterion will prompt an evaluation by a Clinical Center Cardiologist and eligibility will be considered on a case-by-case basis. Should the cardiologist deem the patients findings on work-up to be not clinically significant pathology, the patient will have met this exclusion criterion.

Patients with a history of coronary artery bypass grafting or angioplasty will receive a cardiology evaluation and be considered on a case-by-case basis.

Active hepatitis B or C infection

Human immunodeficiency virus (HIV) seropositive, with positive confirmatory nucleic acid test

Patients known or found to be pregnant.

Patients of childbearing age who are unwilling to practice contraception.

Patients may be excluded at the discretion of the principal investigator (PI)/lead associate investigator (LAI) if it is deemed that allowing participation would represent an unacceptable medical or psychiatric risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-02-22 (Actual); Primary Completion 2014-06-17 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Kanakry, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Alexanian R, Barlogie B, Tucker S. VAD-based regimens as primary treatment for multiple myeloma. Am J Hematol. 1990 Feb;33(2):86-9. doi: 10.1002/ajh.2830330203. PMID 2301376
- [Background] Tosi P, Zamagni E, Cellini C, Plasmati R, Cangini D, Tacchetti P, Perrone G, Pastorelli F, Tura S, Baccarani M, Cavo M. Neurological toxicity of long-term (>1 yr) thalidomide therapy in patients with multiple myeloma. Eur J Haematol. 2005 Mar;74(3):212-6. doi: 10.1111/j.1600-0609.2004.00382.x. PMID 15693790
- [Background] Ogunniyi A, Rodriguez M, Devlin S, Adel N, Landau H, Chung DJ, Lendvai N, Lesokhin A, Koehne G, Mailankody S, Korde N, Reich L, Landgren O, Giralt S, Hassoun H. Upfront use of plerixafor and granulocyte-colony stimulating factor (GCSF) for stem cell mobilization in patients with multiple myeloma: efficacy and analysis of risk factors associated with poor stem cell collection efficiency. Leuk Lymphoma. 2017 May;58(5):1123-1129. doi: 10.1080/10428194.2016.1239261. Epub 2016 Oct 13. PMID 27735212
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-C-0074.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Our study was a relatively small pilot study, with the primary emphasis being on expanding standard stem cell therapy options for patients with multiple myeloma. The plerixafor plus G-CSF combination is used relatively ubiquitously, and several larger studies relating to plerixafor have been performed at large centers that treat multiple myeloma.
Groups:
- Hematopoietic Progenitor Cells (HPC): Subjects will undergo mobilization and collection of HPC, Apheresis for subsequent use in various clinical protocols.
  Filgrastim: Filgrastim will be administered as a single daily dose in a dose range of 10-16ug/kg/day subcutaneously for 5-7days
  Plerixafor: Plerixafor will be given on day 4, 8-10 hours before the day 5 apheresis, dose calculated according to patient weight
  Apheresis: The minimum cluster of differentiation 34 (CD34)+ cell dose that must be collected in order to proceed with a single autologous transplantation is 2 x 10^6 CD34+ cells/kg.
Period: Overall Study
Arm/Group | Hematopoietic Progenitor Cells (HPC)
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hematopoietic Progenitor Cells (HPC): Subjects will undergo mobilization and collection of HPC, Apheresis for subsequent use in various clinical protocols.
  Filgrastim: Filgrastim will be administered as a single daily dose in a dose range of 10-16ug/kg/day subcutaneously for 5-7days
  Plerixafor: Plerixafor will be given on day 4, 8-10 hours before the day 5 apheresis, dose calculated according to patient weight
  Apheresis: The minimum cluster of differentiation 34 (CD34)+ cell dose that must be collected in order to proceed with a single autologous transplantation is 2 x 106^ CD34+ cells/kg.
Arm/Group | Hematopoietic Progenitor Cells (HPC)
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.99 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 48
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving at Least 2 x 10^6 Cluster of Differentiation 34 (CD34) Cells Per Kg Recipient Body Weight on Day 1 of Apheresis
Description: Progenitor cells by apheresis was determined by flow cytometry. The stated goal was a minimum dose of 2x10EE^6/kg following apheresis.
Time Frame: Day 1 of apheresis
Measure: Number; unit: percentage of patients
Arm/Group | Hematopoietic Progenitor Cells (HPC)
Number analyzed (Participants) | 49
percentage of patients | 98

2. Primary Outcome: Percentage of Patients Requiring 2 Days to Achieve at Least 2 x 10^6 Cluster of Differentiation 34 (CD34) Cells Per Kg Recipient Body Weight
Description: Progenitor cells by apheresis was determined by flow cytometry.
Time Frame: Through Day 2 of collection
Measure: Number; unit: percentage of patients
Groups:
- Hematopoietic Progenitor Cells: Subjects will undergo mobilization and collection of HPC, Apheresis for subsequent use in various clinical protocols.
  Filgrastim: Filgrastim will be administered as a single daily dose in a dose range of 10-16ug/kg/day subcutaneously for 5-7days
  Plerixafor: Plerixafor will be given on day 4, 8-10 hours before the day 5 apheresis, dose calculated according to patient weight
  Apheresis: The minimum cluster of differentiation 34 (CD34)+ cell dose that must be collected in order to proceed with a single autologous transplantation is 2 x 106 CD34+ cells/kg.
Arm/Group | Hematopoietic Progenitor Cells
Number analyzed (Participants) | 49
percentage of patients | 2

3. Primary Outcome: Average Number of Cluster of Differentiation 34 (CD34) Cells Collected (Per kg Recipient Body Weight (BW))
Description: Progenitor cells by apheresis was determined by flow cytometry.
Time Frame: Through Day 2 of collection
Measure: Mean (Standard Deviation); unit: Number of CD34 cells per kg/BW (x 10EE6)
Arm/Group | Hematopoietic Progenitor Cells
Number analyzed (Participants) | 49
Number of CD34 cells per kg/BW (x 10EE6) | 6.4 (2.8)

4. Primary Outcome: Median and Standard Deviation of Cluster of Differentiation 34 (CD34) Cells Collected (Per Kg Recipient Body Weight) (BW)
Description: Progenitor cells by apheresis was determined by flow cytometry.
Time Frame: Through Day 2 of collection
Measure: Median (Standard Deviation); unit: Number of CD34 cells per kg/BW (x 10EE6)
Arm/Group | Hematopoietic Progenitor Cells
Number analyzed (Participants) | 49
Number of CD34 cells per kg/BW (x 10EE6) | 6.3 (2.8)

5. Primary Outcome: Range of Cluster of Differentiation 34 (CD34) Cells Collected
Description: Progenitor cells by apheresis was determined by flow cytometry.
Time Frame: Through Day 2 of collection
Measure: Median (Full Range); unit: Number of CD34 cells per kg/BW (x 10EE6)
Arm/Group | Hematopoietic Progenitor Cells
Number analyzed (Participants) | 49
Number of CD34 cells per kg/BW (x 10EE6) | 6.3 [1.7 to 17]

6. Primary Outcome: 25th and 75th Percentile Values of Cluster of Differentiation 34 (CD34) Cells Collected
Description: Progenitor cells by apheresis was determined by flow cytometry.
Time Frame: Through Day 2 of collection
Measure: Number; unit: Number of CD34 cells per kg/BW (x 10EE6)
Arm/Group | Hematopoietic Progenitor Cells
Number analyzed (Participants) | 49
Number of CD34 cells per kg/BW (x 10EE6)
  25th percentile | 4.0
  75th percentile | 8.0

7. Primary Outcome: Number of Hematopoietic Progenitor Cell (HPC) Apheresis Products Collected and Cryopreserved for Subsequent Use in Autologous Hematopoietic Cell Transplantation (AHCT) in Subjects With Plasma Cell Myeloma (PCM)
Description: The cryopreserved stem cells are stored under Good Manufacturing Practice (GMP) conditions in the National Institutes of Health (NIH) Department of Transfusion Medicine until a referring physician requests the products for standard clinical care.
Time Frame: Indefinitely until a referring physician requests the product for standard clinical care or until product(s) is no longer needed and disposed of
Measure: Number; unit: products
Arm/Group | Hematopoietic Progenitor Cells (HPC)
Number analyzed (Participants) | 49
products | 49

8. Secondary Outcome: Number of Participants With Serious and Non-Serious Adverse Events
Description: Here is the number of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: 27 months and 27 days
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Progenitor Cells (HPC)
Number analyzed (Participants) | 49
Participants | 16

9. Secondary Outcome: Percentage of Patients That Required Plerixafor + Granulocyte-colony Stimulating Factor (G-CSF) And Only G-CSF (no Plerixafor)
Description: Percentage of patients that required Plerixafor injection in addition to G-CSF mobilization or none at all
Time Frame: One week of mobilization therapy
Measure: Number; unit: percentage of patients
Arm/Group | Hematopoietic Progenitor Cells
Number analyzed (Participants) | 49
percentage of patients
  Plerixafor + G-CSF | 47
  Only G-CSF (no plerixafor) | 53

10. Secondary Outcome: Percentage of Patients That Achieved or Did Not Achieve 5 x 10^6 Cluster of Differentiation 34 (CD34) Cells/kg
Description: Here is the percentage of patients that achieved or did not achieve 5 x 10^6 CD34 cells/kg in a single apheresis.
Time Frame: Through Day 2 of collection
Measure: Number; unit: percentage of patients
Arm/Group | Hematopoietic Progenitor Cells
Number analyzed (Participants) | 49
percentage of patients
  Achieved 5 x 10EE CD34 cells/kg | 65
  Did not achieve 5 x 10EE CD34 cells/kg | 35

11. Secondary Outcome: Percentage of Patients That Achieved ≥ 2 x 10^6 But Less Than 5 x 10^6 Cluster of Differentiation 34 (CD34) Cells/kg (Day One Collection)
Description: Percentage of patents achieving collecting the minimum but not optimal CD34 cell number.
Time Frame: Day one of collection
Measure: Number; unit: percentage of patients
Arm/Group | Hematopoietic Progenitor Cells
Number analyzed (Participants) | 49
percentage of patients | 31

12. Secondary Outcome: Degree of Tumor Cell Contamination in the Final Product
Description: Flow cytometry to detect tumor contamination.
Time Frame: Day 1 of apheresis
Population: No data from any participant was sufficiently collected to assess tumor cell contamination.
Arm/Group | Hematopoietic Progenitor Cells (HPC)
Number analyzed (Participants) | 0

13. Secondary Outcome: Impact of Plerixafor in the Degree of Tumor Cell Contamination in the Final Product
Description: Flow cytometry to detect tumor contamination.
Time Frame: Day 1 of apheresis
Population: Because no data from any participant was sufficiently collected to assess tumor cell contamination, we were not able to determine the effect of plerixafor on this parameter.
Arm/Group | Hematopoietic Progenitor Cells (HPC)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 27 months and 27 days
Arm/Group | Hematopoietic Progenitor Cells
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 16/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Progenitor Cells (N=49)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1)
Platelet count decreased (Investigations) | 5 (5)

LIMITATIONS AND CAVEATS:
The sample size in outcome measure number 6 was inadequate. Results were not conclusive and the information is determined to be too preliminary to present. No conclusion should be drawn from the reported data for this outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-09-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT01547806/Prot_SAP_ICF_000.pdf